CLINICAL TRIAL: NCT00661622
Title: Immuno-embolization of Hepatic Artery With Granulocyte-macrophage Colony Stimulating Factor (GM-CSF)
Brief Title: Halt Growth of Liver Tumors From Uveal Melanoma With Closure of Liver Artery Following Injection of GM-CSF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04F.445; R21CA103250 (NIH); JT 1280 (Other: JeffTrial Number)
Record Dates: First submitted 2008-04-16; First posted 2008-04-18 (Estimated); Results first posted 2015-06-01 (Estimated); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Uveal Melanoma; Liver Metastases
MeSH Terms: conditions — Uveal Melanoma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Colony-Stimulating Factors; Embolization, Therapeutic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immunoembolization (Experimental): Liver embolization treatment with injection of GM-CSF.
  Interventions: Drug: GM-CSF; Procedure: Embolization
- Plain embolization (Active Comparator): Liver embolization with normal saline injected in place of GM-CSF
  Interventions: Procedure: Embolization

INTERVENTIONS:
Drug: GM-CSF — 2,000 mcg injected into the liver every 4 weeks alternating between right or left lobe when tumors present throughout liver.
  Other Names: granulocyte-macrophage colony stimulating factor
  Arms: Immunoembolization
Procedure: Embolization — A catheter will be introduced to one of the hepatic arteries by way of the femoral artery (groin) to allow injection of GM-CSF in combination with ethiodized oil and gelatin sponge providing a temporary blockage of the blood supply from the hepatic (liver) artery
  Other Names: embo

SUMMARY:
Patients with uveal melanoma metastatic to the liver will be treated with embolization of the hepatic artery every 4 weeks. GM-CSF (granulocyte-macrophage colony simulating factor) or normal saline will be injected into one of the liver arteries with an oily contrast dye, Ethiodol. This is followed by blockage of the artery with small pieces of gelatin sponge (embolization). It is hoped with this novel approach that:

* tumor cells will die due to a loss of their blood supply,
* local inflammatory reactions induced by GM-CSF will kill remaining tumor cells, and
* a systemic immune response against tumor cells may develop.

DETAILED DESCRIPTION:
Patients with uveal melanoma metastatic to the liver will be treated with embolization of the hepatic artery every 4 weeks. GM-CSF (granulocyte-macrophage colony simulating factor) or normal saline will be injected into one of the liver arteries with an oily contrast dye, Ethiodol. This is followed by blockage of the artery with small pieces of gelatin sponge (embolization).

ELIGIBILITY:
Inclusion Criteria:

* Metastatic uveal melanoma in the liver with histological confirmation
* Ability/willingness to give informed consent
* ECOG performance status of 0 or 1
* Adequate renal, liver and bone marrow function

Exclusion Criteria:

* Solitary liver metastasis that is amenable to surgical removal
* Presence of symptomatic liver failure including ascites and hepatic encephalopathy
* Presence of extra-hepatic metastases
* Untreated brain metastases
* Uncontrolled hypertension or congestive heart failure or acute myocardial infarction within 6 months of entry
* Presence of any other medical complication that imply survival of less than six months
* Uncontrolled sever bleeding tendency or active GI bleeding
* Significant allergic reaction to contrast dye or GM-CSF
* Immunosuppressive treatments such as systemic steroids, radiation to pelvis or systemic chemotherapy within 4 weeks
* Previous embolization of the hepatic artery or intrahepatic arterial chemotherapy of liver metastasis
* Active hepatitis with serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) greater than 5 x normal
* HIV infection positive by ELISA
* Pregnancy or breast feeding women
* Biliary obstruction, biliary stent or prior biliary surgery except cholecystectomy
* Significant arteriovenous shunt identified on angiography of the hepatic artery
* Occlusion of main portal vein or inadequate collateral flow around an occluded portal vein

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2004-10; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takami Sato, M.D., Ph.D., Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Plain Embolization: Liver embolization with normal saline injected in place of GM-CSF
  Embolization: A catheter will be introduced to one of the hepatic arteries by way of the femoral artery (groin) to allow injection of normal saline in combination with ethiodized oil and gelatin sponge providing a temporary blockage of the blood supply from the hepatic (liver) artery
Period: Overall Study
Arm/Group | Immunoembolization | Plain Embolization
Started | 26 | 27
Completed | 25 | 27
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immunoembolization | Plain Embolization | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Continuous [Median (Full Range); unit: years] | 56 [28 to 81] | 62 [32 to 90] | 58 [28 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 10 | 15 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 25 | 27 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 27 | 52
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 27 | 52

OUTCOME MEASURES:

1. Primary Outcome: Response of Liver Metastases
Description: Complete response: Disappearance of all target and non-target liver lesions
  Partial response: >= 30% decrease in the sum of the longest diameters (LD) relative to baseline sum LD with at least stable non-target liver lesions
  Stable disease: Absence of change which would qualify as response or progression
  Progression: >= 20% increase in the sum LD in target liver lesions or unequivocal progression of non-target liver lesions in the treated lobe(s) or appearance of one or more new liver lesions >= 10mm in the treated lobe(s)
Time Frame: Every 8 weeks
Measure: Number; unit: participants
Arm/Group | Immunoembolization | Plain Embolization
Number analyzed (Participants) | 26 | 27
participants
  Complete response (CR) | 0 | 0
  Partial response (PR) | 5 | 3
  Stable disease (SD) | 12 | 19
  Progression (PD) | 8 | 5

2. Primary Outcome: Overall Response Rate
Description: Clinical response in the liver metastases will be evaluated after every two embolizations using CT scans or MRI of the abdomen. The sum of the longest diameter (LD) of up to 6 target lesions will be used to determine response. Target indicator lesions will be identified and measured as baseline prior to the first embolization. The same target lesions will then be measured 3 to 4 weeks after every two treatments. The sum of the baseline LDs will be compared to the sum of the LDs after every two treatments.
Time Frame: Baseline then 3 to 4 weeks after every 2 treatments
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Immunoembolization | Plain Embolization
Number analyzed (Participants) | 26 | 27
percentage of participants | 21.2 [10.3 to 30.5] | 16.7 [6.3 to 26.9]

3. Secondary Outcome: Overall Survival
Description: Measured from the start of the treatment to death of patients
Time Frame: Baseline to death
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Immunoembolization | Plain Embolization
Number analyzed (Participants) | 26 | 27
months | 21.5 [18.5 to 24.8] | 17.2 [11.9 to 22.4]

4. Secondary Outcome: Median Progression Free Survival
Description: Measured from the start of the treatment to confirmation of progression of disease by either imaging tests or physical examination.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of one or more new liver lesions >= 10mm in the treated lobe(s).
Time Frame: Baseline to time of progression
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Immunoembolization | Plain Embolization
Number analyzed (Participants) | 26 | 27
months | 3.9 [3.5 to 4.3] | 5.9 [5.5 to 6.2]

5. Secondary Outcome: Systemic Progression Free Survival
Description: as for outcome 4
Time Frame: Baseline to time of progression
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Immunoembolization | Plain Embolization
Number analyzed (Participants) | 26 | 27
months | 10.4 [7.5 to 13.2] | 7.1 [5.0 to 9.1]

ADVERSE EVENTS:
Arm/Group | Immunoembolization | Plain Embolization
Serious Adverse Events (participants affected / at risk) | 3/26 | 5/27
Other Adverse Events (participants affected / at risk) | 26/26 | 23/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunoembolization (N=26) | Plain Embolization (N=27)
Abdominal pain (General disorders) | 0 (0) | 1 (1)
Aneurysms (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Elevated liver enzymes (Hepatobiliary disorders) | 2 (2) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Liver pain (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunoembolization (N=26) | Plain Embolization (N=27)
Agitation (General disorders) | 1 (1) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Anorexia (General disorders) | 4 (6) | 5 (13)
Anxiety (Psychiatric disorders) | 2 (2) | 3 (5)
Athritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Back pain (General disorders) | 0 (0) | 1 (1)
Belching (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bleeding (General disorders) | 1 (2) | 3 (3)
Bleeding at procedure site (General disorders) | 1 (1) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (2) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bruising (Skin and subcutaneous tissue disorders) | 2 (3) | 4 (4)
Bruising at cath site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Burning upper quadrant pain (General disorders) | 0 (0) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Chills/rigors (General disorders) | 4 (6) | 3 (3)
Cold (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (5)
Constipation (Gastrointestinal disorders) | 5 (8) | 5 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Decreased granulocytes (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Decreased hemoglobin (Blood and lymphatic system disorders) | 16 (96) | 17 (147)
Decreased visual acuity (Eye disorders) | 0 (0) | 2 (2)
Decreased WBC (Blood and lymphatic system disorders) | 2 (6) | 4 (4)
Delayed healing of insertion site (General disorders) | 0 (0) | 1 (2)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Diaphoresis (General disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (10) | 5 (8)
Disequilibrium (General disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 3 (3) | 5 (19)
Drug allergy (General disorders) | 0 (0) | 1 (1)
Dry mouth (General disorders) | 0 (0) | 1 (1)
Dysgeusia (General disorders) | 1 (2) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (7) | 2 (2)
Edema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Epigastric pain (General disorders) | 0 (0) | 1 (2)
Fatigue (General disorders) | 11 (26) | 9 (26)
Fever (General disorders) | 9 (15) | 8 (14)
Flatulence (Gastrointestinal disorders) | 2 (3) | 1 (1)
Flu (General disorders) | 1 (1) | 2 (2)
Fluid overload (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Fungal nail infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 4 (10)
Headache (General disorders) | 1 (1) | 3 (6)
Hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Heart palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Hematoma (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hoarseness (General disorders) | 1 (2) | 0 (0)
Hot flashes (General disorders) | 0 (0) | 1 (3)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypertension (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Hypoalbuminemia (Blood and lymphatic system disorders) | 1 (4) | 0 (0)
Hypotension (Blood and lymphatic system disorders) | 3 (6) | 2 (4)
Increased bilirubin (Blood and lymphatic system disorders) | 2 (3) | 2 (2)
Increased alkaline phosphatase (Blood and lymphatic system disorders) | 9 (31) | 9 (36)
Increased creatinine (Blood and lymphatic system disorders) | 2 (8) | 1 (1)
Increased SGOT (Blood and lymphatic system disorders) | 22 (97) | 22 (114)
Increased SGPT (Blood and lymphatic system disorders) | 22 (109) | 22 (117)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Insomnia (General disorders) | 1 (2) | 4 (4)
Irritation (General disorders) | 1 (1) | 0 (0)
Joint pain (General disorders) | 0 (0) | 2 (2)
Lethargy (General disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 8 (32) | 10 (26)
Lymphpenia (Blood and lymphatic system disorders) | 1 (8) | 2 (2)
Muscle cramp (General disorders) | 0 (0) | 1 (1)
Muscle pain (General disorders) | 0 (0) | 1 (1)
Nausea (General disorders) | 17 (63) | 13 (27)
Neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Night sweats (General disorders) | 2 (2) | 1 (2)
Nose bleed (General disorders) | 0 (0) | 2 (3)
Orthostatic hypotension (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 21 (84) | 22 (98)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (11) | 3 (6)
Sensitivity to heat (General disorders) | 1 (1) | 1 (2)
Sinus allergies (General disorders) | 1 (1) | 0 (0)
Sinus pain (General disorders) | 1 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Slurred speech (General disorders) | 1 (1) | 0 (0)
Sprained ankle (General disorders) | 0 (0) | 1 (1)
Stiff neck (General disorders) | 0 (0) | 1 (1)
Sweating (General disorders) | 0 (0) | 2 (4)
Swollen knee (General disorders) | 0 (0) | 1 (1)
Tachycardia (General disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (44) | 5 (13)
Upper respiratory infection (General disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (22) | 6 (9)
Weakness (General disorders) | 0 (0) | 4 (5)
Weight loss (General disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes